CLINICAL TRIAL: NCT03874520
Title: Using Video Transmission for Optimized Telephone Triage of Children With Respiratory Symptoms at the Medical Helpline 1813 in Copenhagen, Denmark
Brief Title: Using Video Transmission for Telephone Triage of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Copenhagen University Hospital at Herlev (Other); Rigshospitalet, Denmark (Other); Copenhagen University Hospital Nordsjælland (Unknown); Copenhagen Academy for Medical Education and Simulation (Other); University of Copenhagen (Other); TrygFonden, Denmark (Industry); Amager-Hvidovre Hospital Research Foundation (Unknown)
Responsible Party: Principal Investigator, Caroline Gren, MD, Emergency Medical Services, Capital Region, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Videotriage 1813
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Telemedicine; Triage; Respiratory Tract Diseases; Pediatrics
Keywords: Telemedicine; Triage; Call Centers; Respiratory Tract Diseases; Pediatrics
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Intervention Model Description: The operators at the medical helpline 1813 will triage children meeting the inclusion criteria using video every other day they are at work, and over telephone the other days. Consequently, the operators are always the same, and the only difference between the two groups of patients will be if video triage or telephone triage is performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video triage (Experimental): The sick child will be assessed on video by the operator at the call-center.
  Interventions: Other: Video triage
- Telephone triage (No Intervention): The sick child will be assessed solely over the telephone by the operator at the call-center.

INTERVENTIONS:
Other: Video triage — The operator will offer the parent calling regarding the sick child to assess the child on video, as compared to the current standard; on the telephone.
  Arms: Video triage

SUMMARY:
Background

The medical helpline 1813 in Copenhagen, Denmark handles telephone calls regarding non-life-threatening medical emergencies. Next to 200,000 calls/year concern children and afterwards about 30% are referred to a pediatric urgent care center. However, most of these children have very mild symptoms, which do neither require treatment nor any tests, but merely parental medical guidance.

Initial assessment; triage, of children on the telephone is difficult, especially when the operator does not know the child or the parents, and when it is difficult to describe the symptoms in medical terms. This may result in both too many not-so-sick children getting unnecessarily referred to hospitals, and perhaps also too few more severely sick children sent to the hospital.

Purpose

This project will study if triage of children by videocalls (video triage) provide greater security for parents and health care personnel in the decision that more children can stay at home after medical guidance, thus causing at least 10% fewer visits to a pediatric urgent care center.

Furthermore, the investigators will study if video triage identifies more children with the need of urgent admission to a Department of Pediatrics.

Method

Children aged 6 months to 5 years with symptoms from the respiratory tract will be triaged by either video or telephone by an operator every other day, in order to compare the results between these two similar groups. In cases of video triage, the parent will receive a text message to their smartphone with a video link.

The safety of video triage will be assessed by reviewing the hospital case reports of all patients for contact within the 48 hours after the 1813 call.

Perspectives

Video assessment at call centers may "give eyes to the operators" and revolutionize telephone triage. The study may result in fewer children referred to hospitals, more appropriate use of resources and better experiences for the families.

DETAILED DESCRIPTION:
Background

Each year the Copenhagen Emergency Services receives approximately 190,000 calls to the medical helpline 1813 regarding sick children younger than 12 years (injuries excluded) (Rasmussen MV, ref. 1). These children are not so sick that the parents call the emergency helpline 112, but the parents need to contact the health care system outside their general practitioners' (GP) opening hours.

After contact with the parents the medical helpline 1813's health professionals have several possibilities for the children; e.g. admitting the children to a Department of Pediatrics, referring them to assessment in Børnelægevagten (a pediatric urgent care center), guiding them to self-care at home, or referring them to their GP the next workday.

Of the 190,000 calls annually regarding sick children, the majority of the calls concerns small children; in 2018, about 175,000 of the calls concerned children younger than 6 years. About 30% of these children were referred to assessment in a pediatric urgent care center. Most of these patients have mild symptoms which do neither require treatment nor paraclinical testing, but merely parental medical guidance. These consultations can be experienced as unnecessary and inappropriate for the sick child and its parents. Moreover, the visits are expensive for the health system.

Telephone triage is difficult, especially when the operator does not know the child or the parents, and when it is difficult to describe symptoms in medical terms. Telemedicine, i.e. the use of communication- and information technology within the healthcare system, is gaining increasing influence in the medical society, also within pediatrics (Olson CA et al, ref. 2). The American Academy of Pediatrics has urged both general pediatricians and pediatric subspecialists to use telemedicine to serve more children (Marcin JP et al, ref. 3).

Two studies both found good agreement between face-to-face and video-assisted assessment of children with respiratory symptoms (Siew L et al, Gattu R et al, ref. 4, 5). Another study about children with acute worsening of asthma, reported that the parents felt safer when the triage of the child was done by a health professional who could watch the child on video, and the health professionals also felt safer with the video triage (Freeman B et al, ref. 6).

Purpose

Does triage of children by videocalls (video triage) provide greater security for parents and health care personnel in the decision that more children can stay at home after medical guidance, thus causing at least 10% fewer visits to Børnelægevagten (a pediatric urgent care center)? Furthermore, doses triage of children by videocalls (video triage) identify more children with the need of urgent admission to a Department of Pediatrics?

The project will investigate the safety of video triage, by subsequently reading in the children's hospital case reports and study if the children have been examined at a pediatric department within the first 48 hours after the 1813 call.

The investigators will also examine the parents' and the operators' experience with the video call, regarding feelings of safety and the technical quality.

The project thus aims to evaluate the value of improving triage with the new technology, video calls.

To our knowledge, there are no other studies of the effect of video calls in the initial triage of children.

Methods

Study design and structure:

The project is a prospective quality improvement study investigating the results of a new intervention.

Initially, a smaller group of nurses is trained in video triage. They will offer video triage every other work day, i.e. one-day video triage and the next day ordinary telephone triage, etc. Consequently, the operators are always the same, and the only difference between the groups will be if video triage is performed.

During the project period, more nurses will be trained in video triage. There will thus be a step-by-step inclusion of nurses who carry out video triage. The project thereby has the character of a stepped wedge randomized trial (Hemming K et al, ref. 7).

The results from video triage days will be compared with results from non-video triage days. The control group will thus be the patients from non-video triage days.

Method of video triage:

Initially 20 operators, all nurses, will be trained in video triage. During the project period, on video days, the operators will offer video triage to children aged 6 months up to and including 5 years, with respiratory symptoms.

The parents will receive a text message with a link on their smartphone, which upon activation starts a video call with the operator at 1813.

The operators will use the medical history as well as the video, i.e. both video and audio, to make a plan for the child together with the parent.

Immediately after the call, the parents will receive a text message with a link to an electronic questionnaire regarding their experience with the call and the assessment of their child.

After the call, the operators at 1813 will also answer an electronic questionnaire, about the experience regarding the call.

On non-video days, the operators will enroll corresponding children to telephone triage. Similarly, these children's parents will receive a text message about their experience with the call, and the nurses will also fill out a questionnaire after these calls.

Within 2 to 8 workdays after the call the project group will read the child's hospital case report, to investigate if the child has been at a hospital within 8 hours or 48 hours after the call to 1813. If the child has been at a hospital, there will be noted for example date, time and diagnosis, and if the child was admitted to an intensive care unit, or in the worst case, got lasting injuries or died.

The data department at the Copenhagen Emergency Services will daily extract data on the children enrolled in the project from a patient treatment database at the Copenhagen Emergency Services, which was established with the approval of the regional information security department. The data sheet will include data on the patient and the call.

Sample size:

In 2018 there were 177,000 calls regarding children up to and including 5 years. Of the 177,000 calls, 9% were referred directly to admission at a department of Pediatrics, 30% were referred to assessment at pediatric urgent care center, 31% were guided in self-care, 25% were advised to call their GPs the next workday and 5% were referred to other options. That is, 56% stayed at home the day the parents called 1813.

The investigators hypothesize that video triage can result in at least 10% more parents staying at home with the child on the day they call 1813, i.e. an increase from 56% to 66%. With a power of 80% and two-sided significance of 95%, a total of 774 children distributed on two equal sized groups of 387 patients should be included according to openepi (http://openepi.com/SampleSize/SSCohort.htm).

If, on the other hand, video triage results in 15% more parents staying at home with the child the day they call 1813, i.e. an increase from 56% to 71%, it is only necessary to include 346 children in total to identify such a difference.

In contrast, if video triage results in 7% more parents staying at home with the child at the day, they call 1813, i.e. an increase from 56% to 63% 1582 children divided into two groups must be included, and if video triage only results in 5% more parents staying at home with the child at the day of the call to 1813, i.e. an increase from 56% to 61% 3102 children divided into two groups must be included. In all cases in according to openepi (http://openepi.com/SampleSize/SSCohort.htm) with a power of 80% and two-sided significance of 95%.

Statistics:

Non-parametric statistics, two-sided and with significance at p-value <0.05.

Interim analyses:

After the first 200 video calls, an interim analysis to study the effect of the video triage will be performed, including the period of time it has taken to enroll these children, as well as how the video triage technically has worked, in order to be able to correct possible problems. The safety will also be reviewed, in order to make sure that the children assessed on video do not have higher admittance rate and/or mortality rate, as a sign that they arrive too late to the hospital.

After the first 400 first calls, another interim analysis to study the effect of video calls will be made. This will also include a study of whether there is a significant difference between the number of children staying at home the day the parents call 1813 using video triage and using common telephone triage.

If no significant difference is revealed the study will go on and the effect of video triage will be evaluated when 774 patients has been enrolled.

If a significant effect is still not revealed between the patients using video triage and using common telephone triage the project will go on until 1600 patients have been included.

If no significant difference is revealed the study will go on and the effect of video triage will be evaluated when 3500 patients has been enrolled. However, the study will not go on more than 6 months.

Perspectives and possible yield

At the end of this initial project, the project group expect to know if use of video triage can increase the number of children who safely can stay at home the day their parents call 1813, i.e. the children are referred to self-care or to their GP. This may be beneficial for the sick child and its parents and there may be a socio-economic win. It will also be known if children with more severe symptoms more often are referred directly to a Department of Pediatrics, rather than to an initial assessment in a pediatric urgent care center.

After the study of the video triage, the management at the Emergency Services Copenhagen can decide if video triage will be an integrated option at the medical helpline 1813.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms presented to the 1813 operator categorized as: coughing/breathing difficulties, cold or suspected influenza.
* Parents are calling from a smartphone with Apple, Windows or Android operating system.

Exclusion Criteria:

* The child has already participated.
* The parent does not call from a Danish telephone number.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 734 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Disposition | disposition is registered by the call operator immediately after the call.
  difference between the two arms in the percentage of children that can stay at home the day the parents call 1813, i.e. referral to self-care or GP, compared to the control group.

SECONDARY OUTCOMES:
Admission | disposition is registered by the call operator immediately after the call.
  difference between the two arms in the percentage of children that are referred to admission at a Department of Pediatrics.
Hospital visits | the hospital chart of all children are read within 2-8 days after the call.
  difference between the two arms in the percentage of how many children that are seen at a hospital within 8 hours or 48 hours after the call to 1813, and does that match the disposition registered by the 1813 nurse? Which diagnosis was given at the hospital?
Safety of disposition choice: percentage of duration of admission | the hospital charts of all children are read within 2-8 days after the call.
  difference between the two arms in the percentage of duration of admission, admission to ICU and mortality.
Nurses' satisfaction: percentage of nurses that were satisfied | the nurses fill out a questionnaire about the call immediately after each call.
  difference between the two arms in the percentage of nurses that were satisfied with the call to a acceptable extent or better in the two groups.
Technical difficulty, nurses | the nurses fill out a questionnaire about the call immediately after each call.
  the number of nurses that found the video call to be technically easy to conduct to a moderate extent or better.
Technical quality of the video call | the nurses fill out a questionnaire about the call immediately after each call.
  the number of nurses that found the sound- and picture quality of the video call as acceptable or better.
Disposition choice | the nurses fill out a questionnaire about the call immediately after each call.
  the percentage of nurses that felt safer about the choice of disposition after video triage compared to after a regular telephone triage, to a acceptable extent or better.
Parents' perception of getting answers to their questions | the parents are sent a link to an online questionnaire immediately after the call to 1813.
  difference between the two arms in the percentage of parents that felt that they got their questions answered during the call to a acceptable extent or better.
Parents' satisfaction about assessment: percentage of parents that felt safe about the assessment | the parents are sent a link to an online questionnaire immediately after the call to 1813.
  difference between the two arms in the percentage of parents that felt safe about the assessment of their children to a acceptable extent or better.
Parents' satisfaction about the plan for the child: percentage of parents that felt safe | the parents are sent a link to an online questionnaire immediately after the call to 1813.
  difference between the two arms in the percentage of parents that felt safe about the plan for their children to a acceptable extent or better
Parents' satisfaction about the call: number of parents in the two arms who were satisfied | the parents are sent a link to an online questionnaire immediately after the call to 1813.
  difference in the number of parents in the two arms who were satisfied with the call to a acceptable extent or better.
Technical difficulty, parents | the parents are sent a link to an online questionnaire immediately after the call to 1813.
  the number of parents that found the video call to be technically easy to conduct to a acceptable extent or better.
Economy | the number of visits to hospitals in each arm will be studied at the completion of enrolling patients.
  how many visits at the pediatric urgent care clinics and at departments of pediatrics, respectively, that could be avoided by using video triage.
Non-participating parents | these parameters will be studied at the completion of enrollment of patients.
  Description of differences in the ages, diagnoses, dispositions between the children whose parents wanted to participate in video triage and those who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Cortes, MD, DrMedSci, Study Chair — Department of Pediatrics, Copenhagen University Hospital Hvidovre
Locations (1):
- Emergency Medical Services, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen, MV. Sektionen for data, controlling og IT, Akutberedskabet, Region Hovedstaden. January 2018 (data extract from the patient database at Emergency Services, Copenhagen)
- [Background] Olson CA, Thomas JF. Telehealth: No Longer an Idea for the Future. Adv Pediatr. 2017 Aug;64(1):347-370. doi: 10.1016/j.yapd.2017.03.009. No abstract available. PMID 28688597
- [Background] COMMITTEE ON PEDIATRIC WORKFORCE; Marcin JP, Rimsza ME, Moskowitz WB. The Use of Telemedicine to Address Access and Physician Workforce Shortages. Pediatrics. 2015 Jul;136(1):202-9. doi: 10.1542/peds.2015-1253. PMID 26122802
- [Background] Siew L, Hsiao A, McCarthy P, Agarwal A, Lee E, Chen L. Reliability of Telemedicine in the Assessment of Seriously Ill Children. Pediatrics. 2016 Mar;137(3):e20150712. doi: 10.1542/peds.2015-0712. Epub 2016 Feb 5. PMID 26908666
- [Background] Gattu R, Scollan J, DeSouza A, Devereaux D, Weaver H, Agthe AG. Telemedicine: A Reliable Tool to Assess the Severity of Respiratory Distress in Children. Hosp Pediatr. 2016 Aug;6(8):476-82. doi: 10.1542/hpeds.2015-0272. PMID 27450148
- [Background] Freeman B, Mayne S, Localio AR, Luberti A, Zorc JJ, Fiks AG. Using Video from Mobile Phones to Improve Pediatric Phone Triage in an Underserved Population. Telemed J E Health. 2017 Feb;23(2):130-136. doi: 10.1089/tmj.2016.0082. Epub 2016 Jun 21. PMID 27328326
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947